CLINICAL TRIAL: NCT07288216
Title: A Phase 2 Posology Study With Long-Term Extension in Participants With Well-Controlled Recurrent Pericarditis to Evaluate the Efficacy and Safety of Transition Regimens to KPL-387 Monotherapy From Standard Therapies
Brief Title: Transition to KPL-387 Monotherapy Dosing & Administration Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kiniksa Pharmaceuticals International, plc (Industry)
Collaborators: Kiniksa Pharmaceuticals, GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KPL-387-C212; 2025-523234-66 (EudraCT Number)
Record Dates: First submitted 2025-12-02; First posted 2025-12-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Pericarditis; Heart Diseases; Pericarditis
Keywords: Recurrence; Recurrent; KPL-387; Recurrent Pericarditis
MeSH Terms: conditions — Pericarditis; Heart Diseases; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Posology KPL-387 (Experimental): In Posology Study, KPL-387 will be administered by subcutaneous (SC) injection through Week 16.
  Interventions: Drug: KPL-387
- Long-Term Extension (Experimental): Participants from Posology Study who continue into the Long-Term Extension will receive KPL-387 for up to 24 months or until KPL-387 is approved for commercial use in that region to treat pericarditis, whichever occurs first.
  Interventions: Drug: KPL-387

INTERVENTIONS:
Drug: KPL-387 — administered by subcutaneous injection

SUMMARY:
The primary objective of this study is to characterize the efficacy and safety of dosing regimens used to transition from prior pericarditis therapies to KPL-387 monotherapy in participants with well-controlled recurrent pericarditis on standard therapies.

DETAILED DESCRIPTION:
During the Posology (Dosing and Administration) Study, participants on oral pericarditis therapies alone (i.e., non-steroidal anti-inflammatory drugs [NSAIDs], colchicine, and/or glucocorticoids) and participants on Interleukin-1 (IL-1) pathway inhibition drugs will transition to KPL-387 per protocol guidelines. Participants will receive KPL-387 for up to 16 weeks in the Posology Study.

At study visits throughout the Posology Study, participants will be queried for symptoms of chest pain (and participants will fill out pericarditis pain numerical rating scale [NRS] scores) and will be assessed for physical signs (e.g., pericardial friction rub) and laboratory evidence of pericarditis activity (e.g., C-reactive protein [CRP]) as well as treatment tolerability and pharmacokinetics (PK). Participants experiencing new or worsening symptoms consistent with pericarditis will be managed per study protocol.

All active, enrolled participants in the Posology Study who have not completed an End of Treatment (EOT) Visit may be eligible to transition into the Long-Term Extension (LTE) following completion of the Week 16 Visit. The Week 16 Visit will serve as both a Posology Study End of Study Visit and a Baseline Visit for the LTE. Participants who choose not to participate in the LTE will complete an EOT Visit followed by a Safety Follow-Up until 8 weeks after the last KPL-387 dose administration.

The open-label LTE is designed to evaluate the long-term efficacy and safety of KPL-387 in recurrent pericarditis (RP). Treatment in the LTE may continue until the participant has received up to 24 months of treatment in the LTE or until KPL-387 is approved for commercial use in that region to treat pericarditis, whichever occurs first.

At study visits throughout the LTE, participants will be queried for symptoms of chest pain (and participants will fill out pericarditis pain NRS scores) and will be assessed for physical signs (e.g., pericardial friction rub) and laboratory evidence of pericarditis activity (e.g., CRP) as well as treatment tolerability and PK. Participants experiencing new or worsening symptoms consistent with pericarditis will be managed as described in the protocol.

ELIGIBILITY:
Key Inclusion Criteria:

* Has well-controlled recurrent pericarditis (i.e., including having CRP < 0.5 mg/dL within 14 days of Baseline and a pericarditis pain NRS score ≤ 3 at Baseline)
* Has a documented history of CRP elevation (> 1 mg/dL) associated with at least one prior acute pericarditis episode, whether the incident event or any pericarditis recurrence
* Has received treatment for RP for at least 3 months prior to Baseline with standard therapy(ies) and is currently on a stable dosing regimen including NSAIDs and/or colchicine, and/or glucocorticoids or an IL-1 pathway inhibitor (anakinra or rilonacept).

Key Exclusion Criteria:

* Has a diagnosis of pericarditis that is secondary to specific prohibited etiologies
* Has had a pericarditis recurrence in the last 3 months prior to Baseline
* Has received an investigational drug during the 4 weeks before study drug administration or is planning to receive an investigational drug at any time during the study.
* Has a history of active or untreated, latent tuberculosis (TB) prior to screening.
* Has a history of immunodeficiency.
* Has a history of immunosuppression, including positive human immunodeficiency virus (HIV) test results.
* Has chest x-ray at Screening or within 12 weeks before first study drug administration, with evidence of malignancy, abnormality consistent with prior or active TB infection or active infection.
* Has a history of malignancy of any organ system within the past 5 years before Screening (other than a successfully treated non-metastatic cutaneous squamous cell carcinoma or basal cell carcinoma and/or localized carcinoma in situ of the cervix).
* Has a known or suspected current active infection or a history of chronic or recurrent infectious disease (> 3 episodes in prior 12 months), including but not limited to, genitourinary infection, chest infection, sinusitis, or skin/soft tissue infection.
* Has had a serious infection, has been admitted to the hospital for an infection, or has been treated for a documented infection requiring antibiotics for a documented infection within 2 weeks prior to first study drug administration.
* Has had an organ transplant (except corneal transplant performed more than 3 months prior to first study drug administration).
* In the Investigator's opinion, has any other medical condition that could adversely affect the subject's participation or interfere with study evaluations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Posology: Proportion of participants free from Pericarditis Recurrence by Week 16 | From first administration of study drug up to Week 16
Long-Term Extension: Annualized rate of Pericarditis Recurrence through the end of the LTE. | Up to 24 Months

SECONDARY OUTCOMES:
Posology: Time to Pericarditis Recurrence by Week 16 | From first administration of study drug up to Week 16
Long Term Extension: Change from LTE Baseline in SF-36v2 Physical Component Summary score through the end of the LTE | Up to 24 Months
  SF-36 (36-item Short Form Survey) Physical Component determines participants' quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; Scores on each item are summed and averaged (range: 0=worst to 100=best) with higher scores indicating better health. Increases from baseline indicate improvement.
Long Term Extension: Change from LTE Baseline in SF-36v2 Mental Component Summary score through the end of the LTE | Up to 24 Months
  SF-36 (36-item Short Form Survey) Mental Component determines participants' quality of life by assessing 1) vitality; 2) limitations in social functioning because of physical or emotional problems; 3) limitations in usual role due to emotional problems; and 4) general mental health. Scores on each item are summed and averaged (range: 0=worst to 100=best) with higher scores indicating better health. Increases from baseline indicate improvement.
Long Term Extension: Change from LTE Baseline in EQ-5D-5L individual index scores over time through the end of the LTE | Up to 24 months
  The EQ-5D-5L (EuroQol-5 Dimension 5-level) is a self-reported health status questionnaire that consists of 6 questions used to calculate a health utility score for use in health economic analysis. There are 2 components to the EQ-5D-5L: a 5-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a visual analogue scale (VAS) that measures health state. Individual and index scores range from 0 to 1, with low scores representing a higher level of dysfunction.
Long Term Extension: Change from LTE Baseline in EQ-5D-5L visual analog scale (VAS) over time through the end of the LTE. | Up to 24 months
  The EQ-5D-5L (EuroQol-5 Dimension 5-level) is a self-reported health status questionnaire that consists of 6 questions used to calculate a health utility score for use in health economic analysis. There are 2 components to the EQ-5D-5L: a 5-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a VAS that measures health state. The VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Investigational Site 002, Santa Monica, California
  - Investigational Site 003, New York, New York
  - Investigational Site 001, Norfolk, Virginia